CLINICAL TRIAL: NCT05955963
Title: Bowel Sounds Analysis in Paediatric Inflammatory Bowel Disease: Relationship With wPCDAI
Acronym: SONO-MICI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2021_843_0018
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Bowel Sounds; Intestinal Inflammation; Crohn Disease
Keywords: bowel sounds; Intestinal Inflammation; Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- paediatric inflammatory bowel disease (Experimental)
  Interventions: Other: Abdominal auscultation

INTERVENTIONS:
Other: Abdominal auscultation — spectral analysis of Bowel sounds

SUMMARY:
The precise and noninvasive evaluation of disease activity among patients with Crohn's disease is not easy, especially for children. It deals with clinical, biological, histological and radiological parameters.

Bowel sounds (BS) when evaluated by a stethoscope are modified by several factors including surgery, infection, drugs or intestinal inflammation. These factors can interact on intestinal motricity. There is a direct relationship between gastrointestinal motility and characteristics of BW. The study of BS using a stethoscope is a simple method, although operator dependent and subjective,with a wide inter and intraindividual variability. Some studies among adults showed interest in the spectral analysis of BS to assess gastrointestinal motility. This more precise and reproducible method is not operator dependent.

To date, no such study has evaluated the correlation between disease activity and the spectral pattern of BS.

of this project is to assess the correlation between disease activity and the spectral pattern of BS in pediatric Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's Disease
* Age between 4 and 17 years
* Follow-up at CHU Amiens-Picardie

Exclusion Criteria:

* Other diseases than Crohn's or treatments affecting the gastrointestinal tract, recent (< 3 months) surgery or refusal to participate (parents or children)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-09-02 (Estimated); Study Completion 2024-06-04 (Estimated)

PRIMARY OUTCOMES:
evaluation of frequency of bowel sounds | one day
evaluation of wPCDAI | one day
  wPCDAI is WEIGHTED PAEDIATRIC CROHN'S DISEASE ACTIVITY INDEX
correlation between wPCDAI and frequency of bowel sounds | one day
  wPCDAI is WEIGHTED PAEDIATRIC CROHN'S DISEASE ACTIVITY INDEX

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No